CLINICAL TRIAL: NCT01304420
Title: Changes in Joint-Cartilage as a Measure of Outcome in Juvenile Idiopathic Arthritis - Assessed by Ultrasonography and Biomarkers
Brief Title: Ultrasonography in Juvenile Idiopathic Arthritis
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 10439
Record Dates: First submitted 2011-01-07; First posted 2011-02-25 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Juvenile Idiopathic Arthritis, Oligoarthritis; Polyarticular Juvenile Rheumatoid Arthritis; Systemic Juvenile Idiopathic Arthritis
Keywords: Juvenile idiopathic arthritis; Ultrasonography; Cartilage; Cartilage biomarkers; Bone biomarkers
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum specimens taken for rutine markers of inflammation.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ultrasonography — Scanning 5 joints bilaterally with an ultrasound scanner
  Other Names: Hitachi EUB-7500

SUMMARY:
The purpose of this study is to analyse the usability of ultrasonography together with biomarkers in the investigation of patients diagnosed with juvenile idiopathic arthritis. The investigators hypothesize that serum and urine markers of cartilage and bone synthesis and degradation, together with ultrasound measurements of joint cartilage thickness, are useful tools in the early evaluation of JIA patients, - as diagnostic, prognostic and monitoring methods.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile idiopathic arthritis: Oligoarticular, polyarticular or systemic onset type.
* Informed consent from parents
* between 5-15 years of age

Exclusion Criteria:

* Other diagnoses that involves bones or cartilage
* Intraarticular steroid injections within 1 month of the trial investigation

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with Juvenile Idiopathic Arthritis, followed in dept of pediatric rheumatology, Aarhus University Hospital, Skejby
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Joint cartilage thickness | 1.5 years
  Joint catilage thickness measured by ultrasonography: knee, ankle, wrist, metacarpophalangeal and proximal interphalangeal joints by MRI: one knee by plain radiographs: knee, ankel and wrist

SECONDARY OUTCOMES:
Level of different biomarkers in serum and urine | 1.5 years
  Level of bone- and cartilage-degradation biomarkers in serum and urine. COMP, CTX-II, RANKL/OPG, PYD/DPD

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric research dept, Aarhus Universityhospital, Skejby, Aarhus, Region Midt, Denmark